CLINICAL TRIAL: NCT03262649
Title: Manitoba Inflammatory Bowel Disease Cohort Study
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: REB#=HS14734 (H2002:040)
Record Dates: First submitted 2017-08-14; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crohn's Disease Cohort: 250 individuals in the Crohn's Disease Cohort
- ulcerative colitis cohort: 108 individuals in the ulcerative colitis cohort

SUMMARY:
The Manitoba Inflammatory Bowel Disease (IBD) Cohort Study participants were drawn from a population-based research registry.

The cohort consisted of 388 adult enrollees with recent IBD onset who completed the baseline survey and interview in 2002 to 2003. Participants were followed every 6 months with surveys and annually with interviews. Diagnosis and disease type were verified by chart review.

DETAILED DESCRIPTION:
The Manitoba Inflammatory Bowel Disease (IBD) Cohort Study, initiated in 2002, is study of adults with IBD who have been tracked prospectively through annual clinical interviews and semiannual surveys. The participants were drawn from a validated population-based research registry, which identified and recruited individuals using an administrative definition of IBD from the comprehensive health data base of Manitoba Health, the single insurer that provides health care to all residents in the province.

The cohort consisted of 388 adult enrollees with recent IBD onset who completed the baseline survey and interview in 2002 to 2003. Participants were followed every 6 months with surveys and annually with interviews. Diagnosis and disease type were verified by chart review. It has been demonstrated that the Cohort is representative of the provincial IBD population as a whole, with comparable age distribution, sex distribution, disease duration, and rural/urban residence.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed within the previous 7 years with Inflammatory Bowel Disease

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Complete data were obtained in the first contact from 388 individuals. Over the first two years of the longitudinal cohort study, there was a modest level of attrition and by the time of the 24 month contact 353 respondents continued to participate.
  The participating persons have been followed annually with in-person interviews and with semi-annual mail-in surveys. By the end of 5 years 353 persons were still participating (a loss of 1.8%/year).
  Participants age was 18-83 and 60% are females. Approximately two thirds live in Winnipeg and the rest live throughout Manitoba including Brandon, Dauphin, Swan River, Flin Flon, Thompson, Winkler and Steinbach. Some subjects live elsewhere in Canada, yet still maintain their participation.
  270 subjects were followed until 2016
Sampling Method: Non-Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2002-03-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Genetic Associations | 2010 to 2016
  Single Nucleotide Variations (SNPs) in gene encoding for membrane transporter proteins were investigated for associations with both IBDs. Target genes included SLC23A1, SLC22A4, SLC22A5, SLC22A23, SLC2A14, SLC2A2 but analyses are not limited to these.

SECONDARY OUTCOMES:
Psychological Functioning 1 | 2010-2014
  The validated 7-item Mastery scale assesses the degree to which persons feel they have some control or mastery over their life to handle day-to-day challenges.
Self Efficacy | 2010-2014
  The IBD- Self Efficacy (SE) is a 29-item scale developed by Keefer et al. (1) based on patient interview, validated self-efficacy measures for other diseases. The instrument assesses the level of confidence in managing various disease-related "tasks," with item scores ranging from 1 (not at all) to 10 (totally), and higher scores reflecting greater disease self-management efficacy. Items were grouped conceptually into 4 subscales, reflecting domains identified by patients with IBD as important [1] managing stress and emotions (sample items: keep from feeling sad; do something to reduce stress); [2] managing medical care (sample items: take medication at instructed times; work out differences with doctors); [3] managing symptoms and disease (sample items: keep diarrhea/urgency from interfering; decrease fatigue); [4] maintaining remission (sample items: engage in self-care; maintain sense of well-being).
Disability | 2010-2014
  The Sheehan Disability Scale is a commonly used and validated instrument that measures disease interference in 3 primary domains of life: work, social, and home, based on a visual analog scale from 0 (no interference) to 10 (very severe interference). (1,2)
  1. Sheehan DV, Harnett-Sheehan K, Raj BA. The measurement of disability. Int Clin Psychopharmacol. 1996;11(suppl 3):89-95.
  2. Leon AC, Olfson M, Portera L, et al. Assessing psychiatric impairment in primary care with the Sheehan Disability Scale. Int J Psychiatry Med. 1997;27:93-105.
Health and Quality of Life 1 | 2010-2014
  Perceived health was assessed using the General Health item from the Medical Outcome Survey Short Form 36, (1) which asks participants to characterize their health in the past year, using 5 response categories from "Excellent" to "Poor."
Disease Activity 1 | 2010-2014
  Current disease activity was assessed using standardized clinical indices, the Harvey-Bradshaw index for CD.
Disease Activity 2 | 2010-2014
  Current disease activity was assessed using standardized clinical indices, the modified Powell-Tuck index for UC.
Disease Activity 3 | 2010-2014
  Recent disease activity was measured with the Manitoba IBD Index
Psychological Functioning 2 | 2010-2014
  The Cohen Perceived Stress Scale is a 14-item questionnaire, with a 5-point Likert response format, that assesses the individual's appraisal of their stress "load" related to chronic and acute stressors.
Psychological Functioning 3 | 2010-2014
  The Brief Symptom Inventory is a well-established measure of current emotional distress related to multiple psychological symptoms, consisting of 53 items.
Psychological Functioning 4 | 2010-2014
  The Psychological Well-being Manifestations Scale consists of 25 items that query 6 general domains of positive experience using a 5-point Likert frequency scale, with higher scores indicating a greater sense of well-being.
Health and Quality of Life 2 | 2010-2014
  The 32-item Inflammatory Bowel Disease Questionnaire is a validated measure that has been extensively used in IBD studies to assess disease-specific quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bernstein, MD, Principal Investigator — University of Mantioba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Benchimol EI, Kaplan GG, Otley AR, Nguyen GC, Underwood FE, Guttmann A, Jones JL, Potter BK, Catley CA, Nugent ZJ, Cui Y, Tanyingoh D, Mojaverian N, Bitton A, Carroll MW, deBruyn J, Dummer TJB, El-Matary W, Griffiths AM, Jacobson K, Kuenzig ME, Leddin D, Lix LM, Mack DR, Murthy SK, Sanchez JNP, Singh H, Targownik LE, Vutcovici M, Bernstein CN. Rural and Urban Residence During Early Life is Associated with Risk of Inflammatory Bowel Disease: A Population-Based Inception and Birth Cohort Study. Am J Gastroenterol. 2017 Sep;112(9):1412-1422. doi: 10.1038/ajg.2017.208. Epub 2017 Jul 25. PMID 28741616
- [Result] Marrie RA, Sellers EAC, Chen H, Fransoo R, Bernstein CN, Hitchon CA, Peschken CA, Garland A. Markedly increased incidence of critical illness in adults with Type 1 diabetes. Diabet Med. 2017 Oct;34(10):1414-1420. doi: 10.1111/dme.13404. Epub 2017 Jul 12. PMID 28626956
- [Result] Restall GJ, Simms AM, Walker JR, Haviva C, Graff LA, Sexton KA, Miller N, Targownik LE, Bernstein CN. Coping with Inflammatory Bowel Disease: Engaging with Information to Inform Health-Related Decision Making in Daily Life. Inflamm Bowel Dis. 2017 Aug;23(8):1247-1256. doi: 10.1097/MIB.0000000000001141. PMID 28498156
- [Result] Singh H, Nugent Z, Yu BN, Lix LM, Targownik LE, Bernstein CN. Higher Incidence of Clostridium difficile Infection Among Individuals With Inflammatory Bowel Disease. Gastroenterology. 2017 Aug;153(2):430-438.e2. doi: 10.1053/j.gastro.2017.04.044. Epub 2017 May 4. PMID 28479377
- [Result] Benchimol EI, Bernstein CN, Bitton A, Carroll MW, Singh H, Otley AR, Vutcovici M, El-Matary W, Nguyen GC, Griffiths AM, Mack DR, Jacobson K, Mojaverian N, Tanyingoh D, Cui Y, Nugent ZJ, Coulombe J, Targownik LE, Jones JL, Leddin D, Murthy SK, Kaplan GG. Trends in Epidemiology of Pediatric Inflammatory Bowel Disease in Canada: Distributed Network Analysis of Multiple Population-Based Provincial Health Administrative Databases. Am J Gastroenterol. 2017 Jul;112(7):1120-1134. doi: 10.1038/ajg.2017.97. Epub 2017 Apr 18. PMID 28417994
- [Result] El-Matary W, Abej E, Deora V, Singh H, Bernstein CN. Impact of Fecal Calprotectin Measurement on Decision-making in Children with Inflammatory Bowel Disease. Front Pediatr. 2017 Jan 25;5:7. doi: 10.3389/fped.2017.00007. eCollection 2017. PMID 28180127
- [Result] Jewel Samadder N, Valentine JF, Guthery S, Singh H, Bernstein CN, Wan Y, Wong J, Boucher K, Pappas L, Rowe K, Bronner M, Ulrich CM, Burt RW, Curtin K, Smith KR. Colorectal Cancer in Inflammatory Bowel Diseases: A Population-Based Study in Utah. Dig Dis Sci. 2017 Aug;62(8):2126-2132. doi: 10.1007/s10620-016-4435-4. Epub 2017 Jan 3. PMID 28050782
- [Result] Nguyen GC, Bernstein CN, Benchimol EI. Risk of Surgery and Mortality in Elderly-onset Inflammatory Bowel Disease: A Population-based Cohort Study. Inflamm Bowel Dis. 2017 Feb;23(2):218-223. doi: 10.1097/MIB.0000000000000993. PMID 27997435
- [Result] Marrie RA, Walker JR, Graff LA, Lix LM, Bolton JM, Nugent Z, Targownik LE, Bernstein CN; CIHR Team "Defining the burden and managing the effects of psychiatric comorbidity in chronic immunoinflammatory disease". Performance of administrative case definitions for depression and anxiety in inflammatory bowel disease. J Psychosom Res. 2016 Oct;89:107-13. doi: 10.1016/j.jpsychores.2016.08.014. Epub 2016 Sep 3. PMID 27663119
- [Result] Graff LA, Sexton KA, Walker JR, Clara I, Targownik LE, Bernstein CN. Validating a Measure of Patient Self-efficacy in Disease Self-management Using a Population-based IBD Cohort: The IBD Self-efficacy Scale. Inflamm Bowel Dis. 2016 Sep;22(9):2165-72. doi: 10.1097/MIB.0000000000000856. PMID 27542132
- [Result] Restall GJ, Simms AM, Walker JR, Graff LA, Sexton KA, Rogala L, Miller N, Haviva C, Targownik LE, Bernstein CN. Understanding Work Experiences of People with Inflammatory Bowel Disease. Inflamm Bowel Dis. 2016 Jul;22(7):1688-97. doi: 10.1097/MIB.0000000000000826. PMID 27271487
- [Result] Bernstein CN, Garland A, Peschken CA, Hitchon CA, Chen H, Fransoo R, Marrie RA. Predictors of ICU Admission and Outcomes 1 Year Post-Admission in Persons with IBD: A Population-based Study. Inflamm Bowel Dis. 2015 Jun;21(6):1341-7. doi: 10.1097/MIB.0000000000000363. PMID 25989339
- [Result] Vagianos K, Clara I, Carr R, Graff LA, Walker JR, Targownik LE, Lix LM, Rogala L, Miller N, Bernstein CN. What Are Adults With Inflammatory Bowel Disease (IBD) Eating? A Closer Look at the Dietary Habits of a Population-Based Canadian IBD Cohort. JPEN J Parenter Enteral Nutr. 2016 Mar;40(3):405-11. doi: 10.1177/0148607114549254. Epub 2014 Sep 4. PMID 25189173
- [Result] Serrano Leon A, Amir Shaghaghi M, Yurkova N, Bernstein CN, El-Gabalawy H, Eck P. Single-nucleotide polymorphisms in SLC22A23 are associated with ulcerative colitis in a Canadian white cohort. Am J Clin Nutr. 2014 Jul;100(1):289-94. doi: 10.3945/ajcn.113.080549. Epub 2014 Apr 16. PMID 24740203
- [Result] Marrie RA, Garland A, Peschken CA, Hitchon CA, Chen H, Fransoo R, Bernstein CN. Increased incidence of critical illness among patients with inflammatory bowel disease: a population-based study. Clin Gastroenterol Hepatol. 2014 Dec;12(12):2063-70.e1-4. doi: 10.1016/j.cgh.2014.03.033. Epub 2014 Apr 12. PMID 24726908
- [Result] Israeli E, Graff LA, Clara I, Walker JR, Lix LM, Targownik LE, Bernstein CN. Low prevalence of disability among patients with inflammatory bowel diseases a decade after diagnosis. Clin Gastroenterol Hepatol. 2014 Aug;12(8):1330-7.e2. doi: 10.1016/j.cgh.2013.12.009. Epub 2013 Dec 17. PMID 24361416
- [Result] Amir Shaghaghi M, Bernstein CN, Serrano Leon A, El-Gabalawy H, Eck P. Polymorphisms in the sodium-dependent ascorbate transporter gene SLC23A1 are associated with susceptibility to Crohn disease. Am J Clin Nutr. 2014 Feb;99(2):378-83. doi: 10.3945/ajcn.113.068015. Epub 2013 Nov 27. PMID 24284447
- [Result] Goldenberg BA, Graff LA, Clara I, Zarychanski R, Walker JR, Carr R, Rogala L, Miller N, Bernstein CN. Is iron deficiency in the absence of anemia associated with fatigue in inflammatory bowel disease? Am J Gastroenterol. 2013 Sep;108(9):1392-7. doi: 10.1038/ajg.2013.14. PMID 24005345
- [Result] Bernstein CN, Ryan JD, Graff LA, Xu W. Commentary: predicting complicated Crohn's disease and surgery--phenotypes, genetics, serology and psychological characteristics of a population-based cohort--authors' reply. Aliment Pharmacol Ther. 2013 Sep;38(5):556-7. doi: 10.1111/apt.12423. No abstract available. PMID 23937465
- [Result] Ryan JD, Silverberg MS, Xu W, Graff LA, Targownik LE, Walker JR, Carr R, Clara I, Miller N, Rogala L, Bernstein CN. Predicting complicated Crohn's disease and surgery: phenotypes, genetics, serology and psychological characteristics of a population-based cohort. Aliment Pharmacol Ther. 2013 Aug;38(3):274-83. doi: 10.1111/apt.12368. Epub 2013 Jun 3. PMID 23725363
- [Result] Bernstein CN, Ng SC, Lakatos PL, Moum B, Loftus EV Jr; Epidemiology and Natural History Task Force of the International Organization of the Study of Inflammatory Bowel Disease. A review of mortality and surgery in ulcerative colitis: milestones of the seriousness of the disease. Inflamm Bowel Dis. 2013 Aug;19(9):2001-10. doi: 10.1097/MIB.0b013e318281f3bb. PMID 23624887
- [Result] Graff LA, Clara I, Walker JR, Lix L, Carr R, Miller N, Rogala L, Bernstein CN. Changes in fatigue over 2 years are associated with activity of inflammatory bowel disease and psychological factors. Clin Gastroenterol Hepatol. 2013 Sep;11(9):1140-6. doi: 10.1016/j.cgh.2013.03.031. Epub 2013 Apr 16. PMID 23602816
- [Result] Targownik LE, Leslie WD, Carr R, Clara I, Miller N, Rogala L, Graff LA, Walker JR, Bernstein CN. Longitudinal change in bone mineral density in a population-based cohort of patients with inflammatory bowel disease. Calcif Tissue Int. 2012 Nov;91(5):356-63. doi: 10.1007/s00223-012-9650-1. Epub 2012 Sep 16. PMID 22983212
- [Result] Wong S, Walker JR, Carr R, Graff LA, Clara I, Promislow S, Rogala L, Miller N, Rawsthorne P, Bernstein CN. The information needs and preferences of persons with longstanding inflammatory bowel disease. Can J Gastroenterol. 2012 Aug;26(8):525-31. doi: 10.1155/2012/735386. PMID 22891177
- [Result] Bernstein MT, Graff LA, Targownik LE, Downing K, Shafer LA, Rawsthorne P, Bernstein CN, Avery L. Gastrointestinal symptoms before and during menses in women with IBD. Aliment Pharmacol Ther. 2012 Jul;36(2):135-44. doi: 10.1111/j.1365-2036.2012.05155.x. Epub 2012 May 24. PMID 22621660
- [Result] Targownik LE, Singh H, Nugent Z, Bernstein CN. The epidemiology of colectomy in ulcerative colitis: results from a population-based cohort. Am J Gastroenterol. 2012 Aug;107(8):1228-35. doi: 10.1038/ajg.2012.127. Epub 2012 May 22. PMID 22613902
- [Result] Shaw SY, Blanchard JF, Bernstein CN. Association between the use of antibiotics and new diagnoses of Crohn's disease and ulcerative colitis. Am J Gastroenterol. 2011 Dec;106(12):2133-42. doi: 10.1038/ajg.2011.304. Epub 2011 Sep 13. PMID 21912437
- [Result] Rawsthorne P, Clara I, Graff LA, Bernstein KI, Carr R, Walker JR, Ediger J, Rogala L, Miller N, Bernstein CN. The Manitoba Inflammatory Bowel Disease Cohort Study: a prospective longitudinal evaluation of the use of complementary and alternative medicine services and products. Gut. 2012 Apr;61(4):521-7. doi: 10.1136/gutjnl-2011-300219. Epub 2011 Aug 11. PMID 21836028
- [Result] Graff LA, Vincent N, Walker JR, Clara I, Carr R, Ediger J, Miller N, Rogala L, Rawsthorne P, Lix L, Bernstein CN. A population-based study of fatigue and sleep difficulties in inflammatory bowel disease. Inflamm Bowel Dis. 2011 Sep;17(9):1882-9. doi: 10.1002/ibd.21580. Epub 2010 Dec 22. PMID 21830266
- [Result] Bernstein CN, El-Gabalawy H, Sargent M, Landers C, Rawsthorne P, Elias B, Targan SR. Assessing inflammatory bowel disease-associated antibodies in Caucasian and First Nations cohorts. Can J Gastroenterol. 2011 May;25(5):269-73. doi: 10.1155/2011/712350. PMID 21647462
- [Result] Longobardi T, Walker JR, Graff LA, Bernstein CN. Health service utilization in IBD: comparison of self-report and administrative data. BMC Health Serv Res. 2011 May 31;11:137. doi: 10.1186/1472-6963-11-137. PMID 21627808
- [Result] Sajobi TT, Lix LM, Clara I, Walker J, Graff LA, Rawsthorne P, Miller N, Rogala L, Carr R, Bernstein CN. Measures of relative importance for health-related quality of life. Qual Life Res. 2012 Feb;21(1):1-11. doi: 10.1007/s11136-011-9914-7. Epub 2011 Apr 24. PMID 21516478
- [Result] Nguyen GC, Nugent Z, Shaw S, Bernstein CN. Outcomes of patients with Crohn's disease improved from 1988 to 2008 and were associated with increased specialist care. Gastroenterology. 2011 Jul;141(1):90-7. doi: 10.1053/j.gastro.2011.03.050. Epub 2011 Mar 31. PMID 21458455
- [Result] Bernstein CN, Nugent Z, Blanchard JF. 5-aminosalicylate is not chemoprophylactic for colorectal cancer in IBD: a population based study. Am J Gastroenterol. 2011 Apr;106(4):731-6. doi: 10.1038/ajg.2011.50. Epub 2011 Mar 15. PMID 21407180
- [Result] Singh H, Nugent Z, Demers AA, Kliewer EV, Mahmud SM, Bernstein CN. The reduction in colorectal cancer mortality after colonoscopy varies by site of the cancer. Gastroenterology. 2010 Oct;139(4):1128-37. doi: 10.1053/j.gastro.2010.06.052. Epub 2010 Jun 20. PMID 20600026
- [Result] Nugent Z, Blanchard JF, Bernstein CN. A population-based study of health-care resource use among infliximab users. Am J Gastroenterol. 2010 Sep;105(9):2009-16. doi: 10.1038/ajg.2010.139. Epub 2010 Apr 6. PMID 20372114
- [Result] Graff LA, Walker JR, Clara I, Lix L, Miller N, Rogala L, Rawsthorne P, Bernstein CN. Stress coping, distress, and health perceptions in inflammatory bowel disease and community controls. Am J Gastroenterol. 2009 Dec;104(12):2959-69. doi: 10.1038/ajg.2009.529. Epub 2009 Sep 15. PMID 19755973
- [Result] Clara I, Lix LM, Walker JR, Graff LA, Miller N, Rogala L, Rawsthorne P, Bernstein CN. The Manitoba IBD Index: evidence for a new and simple indicator of IBD activity. Am J Gastroenterol. 2009 Jul;104(7):1754-63. doi: 10.1038/ajg.2009.197. Epub 2009 May 19. PMID 19455122
- [Result] Singh S, Graff LA, Bernstein CN. Do NSAIDs, antibiotics, infections, or stress trigger flares in IBD? Am J Gastroenterol. 2009 May;104(5):1298-313; quiz 1314. doi: 10.1038/ajg.2009.15. Epub 2009 Mar 31. PMID 19337242
- [Result] Stainier DY, Bilder DH, Gilbert W. Spatial domains in the developing forebrain: developmental regulation of a restricted cell surface protein. Dev Biol. 1991 Sep;147(1):22-31. doi: 10.1016/s0012-1606(05)80004-1. PMID 1879609
- [Result] Leslie WD, Miller N, Rogala L, Bernstein CN. Body mass and composition affect bone density in recently diagnosed inflammatory bowel disease: the Manitoba IBD Cohort Study. Inflamm Bowel Dis. 2009 Jan;15(1):39-46. doi: 10.1002/ibd.20541. PMID 18623166
- [Result] Okazaki T, Wang MH, Rawsthorne P, Sargent M, Datta LW, Shugart YY, Bernstein CN, Brant SR. Contributions of IBD5, IL23R, ATG16L1, and NOD2 to Crohn's disease risk in a population-based case-control study: evidence of gene-gene interactions. Inflamm Bowel Dis. 2008 Nov;14(11):1528-41. doi: 10.1002/ibd.20512. PMID 18521914
- [Result] Lix LM, Graff LA, Walker JR, Clara I, Rawsthorne P, Rogala L, Miller N, Ediger J, Pretorius T, Bernstein CN. Longitudinal study of quality of life and psychological functioning for active, fluctuating, and inactive disease patterns in inflammatory bowel disease. Inflamm Bowel Dis. 2008 Nov;14(11):1575-84. doi: 10.1002/ibd.20511. PMID 18512245
- [Result] Leslie WD, Miller N, Rogala L, Bernstein CN. Vitamin D status and bone density in recently diagnosed inflammatory bowel disease: the Manitoba IBD Cohort Study. Am J Gastroenterol. 2008 Jun;103(6):1451-9. doi: 10.1111/j.1572-0241.2007.01753.x. Epub 2008 Apr 16. PMID 18422819
- [Result] Rogala L, Miller N, Graff LA, Rawsthorne P, Clara I, Walker JR, Lix L, Ediger JP, McPhail C, Bernstein CN. Population-based controlled study of social support, self-perceived stress, activity and work issues, and access to health care in inflammatory bowel disease. Inflamm Bowel Dis. 2008 Apr;14(4):526-35. doi: 10.1002/ibd.20353. PMID 18183608
- [Result] Bernstein CN, Wajda A, Blanchard JF. The incidence of arterial thromboembolic diseases in inflammatory bowel disease: a population-based study. Clin Gastroenterol Hepatol. 2008 Jan;6(1):41-5. doi: 10.1016/j.cgh.2007.09.016. Epub 2007 Dec 11. PMID 18063423
- [Result] Ediger JP, Walker JR, Graff L, Lix L, Clara I, Rawsthorne P, Rogala L, Miller N, McPhail C, Deering K, Bernstein CN. Predictors of medication adherence in inflammatory bowel disease. Am J Gastroenterol. 2007 Jul;102(7):1417-26. doi: 10.1111/j.1572-0241.2007.01212.x. Epub 2007 Apr 16. PMID 17437505
- [Result] Graff LA, Walker JR, Lix L, Clara I, Rawsthorne P, Rogala L, Miller N, Jakul L, McPhail C, Ediger J, Bernstein CN. The relationship of inflammatory bowel disease type and activity to psychological functioning and quality of life. Clin Gastroenterol Hepatol. 2006 Dec;4(12):1491-1501. doi: 10.1016/j.cgh.2006.09.027. PMID 17162241
- [Result] Brant SR, Wang MH, Rawsthorne P, Sargent M, Datta LW, Nouvet F, Shugart YY, Bernstein CN. A population-based case-control study of CARD15 and other risk factors in Crohn's disease and ulcerative colitis. Am J Gastroenterol. 2007 Feb;102(2):313-23. doi: 10.1111/j.1572-0241.2006.00926.x. Epub 2006 Nov 13. PMID 17100976
- [Result] Tang LY, Rawsthorne P, Bernstein CN. Are perineal and luminal fistulas associated in Crohn's disease? A population-based study. Clin Gastroenterol Hepatol. 2006 Sep;4(9):1130-4. doi: 10.1016/j.cgh.2006.06.021. Epub 2006 Aug 14. PMID 16905369
- [Result] Longobardi T, Bernstein CN. Health care resource utilization in inflammatory bowel disease. Clin Gastroenterol Hepatol. 2006 Jun;4(6):731-43. doi: 10.1016/j.cgh.2006.02.013. Epub 2006 May 2. PMID 16631415
- [Result] Burgmann T, Clara I, Graff L, Walker J, Lix L, Rawsthorne P, McPhail C, Rogala L, Miller N, Bernstein CN. The Manitoba Inflammatory Bowel Disease Cohort Study: prolonged symptoms before diagnosis--how much is irritable bowel syndrome? Clin Gastroenterol Hepatol. 2006 May;4(5):614-20. doi: 10.1016/j.cgh.2006.03.003. Epub 2006 Apr 17. PMID 16630762
- [Result] Bernstein CN, Wajda A, Blanchard JF. The clustering of other chronic inflammatory diseases in inflammatory bowel disease: a population-based study. Gastroenterology. 2005 Sep;129(3):827-36. doi: 10.1053/j.gastro.2005.06.021. PMID 16143122
- [Result] Goldenberg BA, Rawsthorne P, Bernstein CN. The utility of 6-thioguanine metabolite levels in managing patients with inflammatory bowel disease. Am J Gastroenterol. 2004 Sep;99(9):1744-8. doi: 10.1111/j.1572-0241.2004.30415.x. PMID 15330913
- [Result] Bernstein CN, Bector S, Leslie WD. Lack of relationship of calcium and vitamin D intake to bone mineral density in premenopausal women with inflammatory bowel disease. Am J Gastroenterol. 2003 Nov;98(11):2468-73. doi: 10.1111/j.1572-0241.2003.07676.x. PMID 14638350
- [Result] Bernstein CN, Leslie WD, Taback SP. Bone density in a population-based cohort of premenopausal adult women with early onset inflammatory bowel disease. Am J Gastroenterol. 2003 May;98(5):1094-100. doi: 10.1111/j.1572-0241.2003.07415.x. PMID 12809833
- [Result] Bernstein CN, Blanchard JF, Rawsthorne P, Yu N. The prevalence of extraintestinal diseases in inflammatory bowel disease: a population-based study. Am J Gastroenterol. 2001 Apr;96(4):1116-22. doi: 10.1111/j.1572-0241.2001.03756.x. PMID 11316157
- [Result] Bernstein CN, Blanchard JF, Houston DS, Wajda A. The incidence of deep venous thrombosis and pulmonary embolism among patients with inflammatory bowel disease: a population-based cohort study. Thromb Haemost. 2001 Mar;85(3):430-4. PMID 11307809
- [Result] Bernstein CN, Blanchard JF, Leslie W, Wajda A, Yu BN. The incidence of fracture among patients with inflammatory bowel disease. A population-based cohort study. Ann Intern Med. 2000 Nov 21;133(10):795-9. doi: 10.7326/0003-4819-133-10-200011210-00012. PMID 11085842
- [Derived] Amir Shaghaghi M, Zhouyao H, Tu H, El-Gabalawy H, Crow GH, Levine M, Bernstein CN, Eck P. The SLC2A14 gene, encoding the novel glucose/dehydroascorbate transporter GLUT14, is associated with inflammatory bowel disease. Am J Clin Nutr. 2017 Dec;106(6):1508-1513. doi: 10.3945/ajcn.116.147603. Epub 2017 Sep 27. PMID 28971850